CLINICAL TRIAL: NCT01143259
Title: A Randomized, Double Blind, Placebo Controlled Study to Study Intermountain Healthcare's Enhanced Recovery Protocol for Colon Surgery With and Without Alvimopan Use
Brief Title: Intermountain Healthcare's Enhanced Recovery Protocol for Colon Surgery With and Without Alvimopan Use
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Intermountain Health Care, Inc. (Other)
Collaborators: Cubist Pharmaceuticals LLC, a subsidiary of Merck & Co., Inc. (Rahway, New Jersey USA) (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: Intermountain Alvimopan1017978
Record Dates: First submitted 2010-05-24; First posted 2010-06-14 (Estimated); Results first posted 2014-05-19 (Estimated); Last update posted 2014-09-04 (Estimated); Status verified 2014-04

CONDITIONS: Ileus
Keywords: Ileus; Post operative ileus
MeSH Terms: conditions — Ileus | interventions — alvimopan; Polyethylene

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- 300 mg Polyethylene (Placebo Comparator)
  Interventions: Drug: 300 mg Polyethylene
- Alvimopan (Active Comparator)
  Interventions: Drug: Alvimopam

INTERVENTIONS:
Drug: Alvimopam — The treatment group will receive 12mg of Alvimopan by mouth 30 to 90 minutes before surgery and twice daily till discharge or to a maximum of 7 days (15 doses, total) after surgery.12 mg by mouth 30 to 90 minutes before surgery and twice daily till discharge or to a maximum of 7 days.
  Other Names: Entereg
  Arms: Alvimopan
Drug: 300 mg Polyethylene — The control group will receive 300mg of polyethylene glyco by mouth 30 to 90 minutes before surgery and twice daily till discharge or to a maximum of 7 days (15 doses, total) after surgery.
  Arms: 300 mg Polyethylene

SUMMARY:
The purpose of this study is to determine if the addition of alvimopan to our care process model for colon resection patients will decrease length of stay. The care process model is a combination of optimal IV fluid management, early feeding, early ambulation, patient education, and pain management.

DETAILED DESCRIPTION:
Narcotic pain medicines bind mu-opioid receptors in the bowel and delay the return of normal function. Alvimopan is a peripherally acting mu-opioid receptor antagonist that blocks mu-opioid receptors in the gastrointestinal tract but does not compromise central nervous system-mediated opioid-based analgesia. Length of stay is an important surrogate measure of quality after colon surgery and the most common reason for prolonged Length of Stay after abdominal surgery is delayed gastrointestinal recovery (postoperative ileus).

The Food and Drug Administration has approved alvimopan (dosed preoperatively and twice daily postoperatively for up to 15 in-hospital doses) for the acceleration of upper and lower gastrointestinal recovery after partial bowel resection with primary anastomosis. In the 5 phase III alvimopan efficacy trials, a simple standardized accelerated postoperative care pathway was used rather than a comprehensive, multidisciplinary colon surgery care process model that is used by Intermountain Healthcare. In the most recently completed alvimopan phase III trial, the mean postoperative length of stay was 5.2 days whereas the mean length of stay at Intermountain Healthcare is 4.4 days without the addition of alvimopan to the multidisciplinary colon care process model.

This trial will investigate if the addition of alvimopan to the Intermountain Healthcare multidisciplinary care process can decrease length of stay compared with the multidisciplinary care process plus placebo.

ELIGIBILITY:
Inclusion Criteria:

1. Age > 18
2. Patient scheduled to receive opioid-based postoperative pain management ≥ 48 hrs
3. Elective colon/rectal resection with anastomosis as primary procedure
4. Patient enrolled in multidisciplinary colon care process

Exclusion Criteria:

1. Pregnancy or lactation
2. Chronic opioid use or > 3 doses in 7 days prior to surgery
3. History of multiple previous abdominal operations, gastrectomy, bariatric surgery, short bowel syndrome
4. Complete bowel obstruction
5. Patients with end-stage renal disease as defined by the need for dialysis and the commonly accepted threshold for dialysis is a Glomerular Filtration Rate of < 15.
6. Patients with severe hepatic impairment (Childs-Pugh class C)
7. ASA 4 or 5 (ASA 4 s incapacitating systemic disease that is a constant threat to life)
8. Non-English speaking patients

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 274 (Actual)
Dates: Start 2010-05; Primary Completion 2012-06 (Actual); Study Completion 2012-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Bob Moesinger, MD, Principal Investigator — Intermountain Health Care, Inc.; Matthew Peters, RN, Study Director — Intermountain Health Care, Inc.
Locations (9):
- United States (9):
  - American Fork Hospital, American Fork, Utah
  - Valley View Hospital, Cedar City, Utah
  - Logan Regional Hospital, Logan, Utah
  - Intermoutain Medical Center, Murray, Utah
  - McKay-Dee Hospital, Ogden, Utah
  - Utah Valley, Provo, Utah
  - LDS Hospital, Salt Lake City, Utah
  - Alta View Hospital, Sandy City, Utah
  - Dixie Regional, St. George, Utah

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Date of first enrollment5-24-2010 Date of last enrollment 6-13-2012 Patients were identified in surgeons office and then screen by study coordinators for eligibility.
Pre-assignment Details: Most common exclusion were patients with history of opioid us > 3 doses in 7 days prior to surgery.
Groups:
- 300 mg Polyethylene: Control Group : The control group will receive 300mg of polyethylene glyco by mouth 30 to 90 minutes before surgery and twice daily till discharge or to a maximum of 7 days (15 doses, total) after surgery.
- Alvimopan: Treatment Group : The treatment group will receive 12mg of Alvimopan by mouth 30 to 90 minutes before surgery and twice daily till discharge or to a maximum of 7 days (15 doses, total) after surgery.12 mg by mouth 30 to 90 minutes before surgery and twice daily till discharge or to a maximum of 7 days.
Period: Overall Study
Arm/Group | 300 mg Polyethylene | Alvimopan
Started | 136 | 138
Completed | 113 | 118
Not Completed | 23 | 20
Not completed — Withdrawal by Subject | 3 | 2
Not completed — Protocol Violation | 13 | 9
Not completed — Screen Failure | 7 | 9

BASELINE CHARACTERISTICS:
Groups:
- 300 mg Polyethylene: Control Group: The control group will receive 300mg of polyethylene glyco by mouth 30 to 300 minutes before surgery and twice daily till discharge or to a maximum of 7 days (15 doses, total) after surgery.
- Alvimopan: Treatment Group: The treatment group will receive 12mg of Alvimopan by mouth 30 to 300 minutes before surgery and twice daily till discharge or to a maximum of 7 days (15 doses, total) after surgery.12 mg by mouth 30 to 90 minutes before surgery and twice daily till discharge or to a maximum of 7 days.
- Total: Total of all reporting groups
Arm/Group | 300 mg Polyethylene | Alvimopan | Total
Number analyzed (Participants) | 136 | 138 | 274
Age, Customized [Mean (Full Range); unit: years]
  Age | 61 [20 to 89] | 61 [18 to 87] | 61 [18 to 89]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 66 | 69 | 135
  Male | 70 | 69 | 139
Region of Enrollment [Number; unit: participants]
  United States | 136 | 138 | 274
Mean BMI [Median (Full Range); unit: Kg/M^2] | 28 [16 to 60] | 29 [19 to 51] | 28 [16 to 60]
Total Cases Using An Open Approach [Number; unit: Cases] — This only includes those surgical cases that were used in the analysis of the study which had surgery with an open approach versus laparoscopic.
  Cases | 43 | 25 | 68

OUTCOME MEASURES:

1. Primary Outcome: Measure of Improvement Over the Standard
Description: Determine if alvimopan addition to the multidisciplinary care process will result in decreased length of stay compared with the multidisciplinary care process plus placebo. Length of stay is determined by how many days a patient stays in the hospital. This is calculated by subtracting the discharge date from the admit date.
Time Frame: Number of days the patient stayed in the hospital [Time frame: Inpatient admit day to discharge day]
Population: The overall baseline number of participants is 274. The total number of participants that were included in the study was 248. There were 26 participants that either chose to not participate in the study after starting, or had protocol violations that excluded them from being included in the measured population.
Measure: Mean (Full Range); unit: Days in the hospital
Arm/Group | 300 mg Polyethylene | Alvimopan
Number analyzed (Participants) | 125 | 123
Days in the hospital | 4.97 [1.9 to 30.2] | 3.98 [1.2 to 28.2]

2. Secondary Outcome: Hospital Cost
Description: Total Cost of hospital stay inflation adjusted to 2010 dollars.
Time Frame: Upon discharge
Population: as for outcome 1
Measure: Mean (Full Range); unit: Dollars
Arm/Group | 300 mg Polyethylene | Alvimopan
Number analyzed (Participants) | 125 | 123
Dollars | 14,520 [6170 to 78,521] | 12,834 [5,788 to 78,708]

ADVERSE EVENTS:
Time Frame: 30 Days after hospital discharge
Groups:
- Alvimopan: Treatment Group: The treatment group will receive 12mg of Alvimopan by mouth 30 to 300 minutes before surgery and twice daily till discharge or to a maximum of 7 days (15 doses, total) after surgery.
Arm/Group | 300 mg Polyethylene | Alvimopan
Serious Adverse Events (participants affected / at risk) | 0/136 | 0/138
Other Adverse Events (participants affected / at risk) | 13/136 | 3/138
OTHER ADVERSE EVENTS (reported when occurring in more than 2% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | 300 mg Polyethylene (N=136) | Alvimopan (N=138)
Post Operative Ileus (Gastrointestinal disorders) | 13 (13) | 3 (3) — National Surgical Quality Improvement Project definition-presence of nasogastric tube or order for nothing by mouth > postoperative day 4)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No